CLINICAL TRIAL: NCT00543036
Title: Efficacy and Safety of the Hcoil Deep TMS for the Treatment of Cannabis Addiction
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shalvata Mental Health Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SH 30107
Record Dates: First submitted 2007-10-11; First posted 2007-10-12 (Estimated); Last update posted 2007-10-12 (Estimated); Status verified 2007-08

CONDITIONS: Marijuana Abuse
Keywords: Cannabis; Addiction; Craving; TMS
MeSH Terms: conditions — Marijuana Abuse; Behavior, Addictive

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Device: H-Coil deep TMS

SUMMARY:
Evaluation of efficacy and safety of H-coil deep transcranial magnetic stimulation 9 week treatment trial for cannabis addiction as assessed by measures of drug intake and craving.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female, aged 21-70 years, who meet DSM-IV TR diagnostic criteria for cannabis abuse and are motivated to quit cannabis use as assessed in the screening visit and gave their written informed consent to participate in the study.

Exclusion Criteria:

* History of a primary major psychiatric other then cannabis abuse, or cognitive disorder according to DSM-IV TR criteria.
* Hamilton depression scale rated 25 and above (moderate to severe depression)
* Current alcohol or other substance abuse or dependence
* Alcohol or other substance abuse or dependence during the last 12 months before recruitment.
* History of or evidence of significant brain malformation,neoplasm, head injury, cerebral vascular events,neurodegenerative disorder or brain surgery.
* Severe somatic co-morbidity
* History of seizures Cardiac pace maker or other electronic implants Pregnancy and lactation

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Ziv Carmel, M.D, Principal Investigator — Shalvata MHC affiliated to Tel-Aviv universtiy, Sackler school of medicine; Abraham Zangen, Ph.D., Principal Investigator — Weizmann Institute, Rehovot, Israel
Locations (1):
- Shalvata Mental Health Center, Hod HaSharon, Israel